CLINICAL TRIAL: NCT01577888
Title: Safety and Feasibility Study of the Shockwave Lithoplasty System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TD-0047
Record Dates: First submitted 2012-04-11; First posted 2012-04-16 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Vascular Disease
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lithotripsy Treatment (Experimental): Shockwave System Treatment -Lithotripsy-enhanced, low-pressure balloon dilation of calcified, stenotic peripheral arteries.
  Interventions: Device: Shockwave System Treatment

INTERVENTIONS:
Device: Shockwave System Treatment — Shockwave System Treatment during vascular disease intervention.

SUMMARY:
To study the early safety and performance of the Shockwave Medical System in subjects to demonstrate that the device can safely and effectively deliver localized energy for the treatment of vascular disease.

DETAILED DESCRIPTION:
Shockwave Medical, Inc. intends to conduct a prospective, single-arm, single-center, First in Human study designed to evaluate the early safety and feasibility of the Shockwave Lithoplasty System in subjects with heavily calcified infrainguinal arteries with 3.75mm to 6mm reference vessel diameter at target site. The Shockwave Lithoplasty System is indicated to generate sonic shockwave energy within the target treatment site and disrupt calcium within the lesion to allow for subsequent dilation of a peripheral artery stenosis using low balloon pressure. Up to 10 subjects will be enrolled to undergo lihtoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Patient or patient's legal representative have been informed of the nature of the study, agrees to participate and has signed the approved consent form.
* Female subjects of childbearing potential have a negative pregnancy test less than 7 days before the procedure.
* Patient is able and willing to comply with all assessments in the study.
* Peripheral arterial disease of Rutherford Category 2, 3, 4, and 5.
* Ability to tolerate an antiplatelet agent (i.e. aspirin, clopidigrel or prasagrel).
* Meets Angiographic Inclusion Criteria

Exclusion Criteria:

* Patients with peripheral arterial disease of Rutherford Category 6.
* Severe or infected gangrene of the lower extremity.
* Planned major amputation.
* Previously implanted stent at the treatment site.
* Patient with an externally-connected intracardiac catheter or pacemaker.
* Patient with an implantable pacemaker or defibrillator.
* Patient has connective tissue disease (e.g., Marfan's syndrome).
* Patient has a hypercoagulable disorder.
* Patient has allergy to imaging contrast media for which they cannot be premedicated.
* Patient is in acute renal failure or chronic renal insufficiency or failure as measured by a serum creatinine of >19.5 µmol/L.
* Patient has active systemic infection.
* Patient has less than a one year life expectancy.
* Patient is pregnant or nursing.
* Patient is participating in another research study involving an investigational agent that has not reached the primary endpoint.
* Patient has other medical, social or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment, and the procedures and evaluations pre- and post-treatment.
* Chronic total occlusion of target vessel.
* Chronic total occlusion of inflow vessel.
* Highly tortuous arteries (bends greater than 30 degrees over the arc length of the balloon)
* Patients requiring concurrent intervention below the most distal target lesion.
* Inflow disease: Stenosis of >50% in vessel proximal to the target lesion which requires treatment with Drug Eluting Balloon (DEB) or atherectomy.
* Prior procedure in target leg within past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Safety determined by 30day New-Onset Serious Adverse Events | 30 day
  New Onset Serious Adverse Events (SAE) include death, device-related surgery or repeat hospitalization, occlusion, or major unplanned amputation through 30 days following the procedure.

SECONDARY OUTCOMES:
Angiographic Success as measured by residual stenosis <30% reference vessel. | Peri-Procedural

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Holden, MD, Principal Investigator — Auckland City Hospital
Locations (1):
- Auckland City Hospital, Auckland, New Zealand